CLINICAL TRIAL: NCT06816953
Title: Cartilage Biomarkers and HEAD-US Score in Severe Hemophilia A Patients Receiving Low Dose FVIII Prophylaxis
Brief Title: Cartilage Biomarkers and HEAD-US Score in Severe Hemophilia A Patients Receiving FVIII Prophylaxis
Acronym: HEADUS_SHA8
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0736/67; Ratchadapisek Research Fund (Other Grant/Funding Number: Chulalongkorn University)
Record Dates: First submitted 2025-01-19; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia A
Keywords: Hemophilic arthropathy; Diagnostic ultrasound; Severe hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Intervention Model Description: PwSHA receiving low-dose FVIII prophylaxis for ≥6 months were enrolled. Weight-based low-dose FVIII prophylaxis (10-15 IU/kg, 1-3 times/week) was continued for 4 months, then switched to PK-guided low-dose EHL FVIII prophylaxis, targeting a trough FVIII activity of 1 IU/dL, for another 4 months. ESR, CRP, ferritin, and CTX-II were measured at week 8 (during the weight-based low-dose regimen) and at week 24 (during the PK-guided regimen). HEAD-US scores were also compared at weeks 16 and 32. Bleeding rates and quality-of-life (QoL) score were analyzed parallelly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard low dose FVIII prophylaxis (Experimental): Standard weight based low dose FVIII concentrates prophylaxis
  Interventions: Diagnostic Test: HEAD-US; Diagnostic Test: Urinary carboxy-terminal cross linked telopeptide of type II collagen; Diagnostic Test: Inflammatory markers
- PK guided Extended half life FVIII prophylaxis (Active Comparator): Pharmacokinetic guided extended half life FVIII prophylaxis
  Interventions: Diagnostic Test: HEAD-US; Diagnostic Test: Urinary carboxy-terminal cross linked telopeptide of type II collagen; Diagnostic Test: Inflammatory markers

INTERVENTIONS:
Diagnostic Test: HEAD-US — HEAD-US for evaluate haemophilic arthropathy in 6 joints. (Elbow, Knee, Ankle)
Diagnostic Test: Urinary carboxy-terminal cross linked telopeptide of type II collagen — Cartilage biomarker represent cartilage degradation
Diagnostic Test: Inflammatory markers — Inflammatory markers included CBC, Ferritin, ESR, CRP

SUMMARY:
Patients with severe hemophilia A often develop joint complication requiring careful monitoring. This study aimed to compare the effectiveness of standard low dose weight-based FVIII concentrates (CFCs) prophylaxis with pharmacokinetic-guided extended half-life FVIII concentrates (eHLFVIII) using cartilage biomarkers and HEAD-US score.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe hemophilia A
* previously receiving standard low dose FVIII prophylaxis 1-3 times per week for at least 6 months prior to enrollment in the project
* no history of FVIII inhibitor (<0.6 Bethesda unit/ml)
* obtained consent from both patients and their parents

Exclusion Criteria:

* patients with underlying condition affecting the joints such as osteoarthritis, metabolic bone disease, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of standard low dose FVIII concentrate prophylaxis and PK-guided eHL FVIII prophylaxis | From enrollment to the end of treatment at 32 weeks
  To compare the effectiveness of standard weight base FVIII concentrate prophylaxis and pharmacokinetic guided extended half life FVIII prophylaxis in managing hemophilic arthropathy using cartilage biomarkers.
The effectiveness of standard low dose FVIII concentrate prophylaxis and PK-guided eHL FVIII prophylaxis | From enrollment to the end of treatment at 32 weeks
  To compare the effectiveness of standard weight base FVIII concentrate prophylaxis and pharmacokinetic guided extended half life FVIII prophylaxis in managing hemophilic arthropathy using HEAD-US score.

SECONDARY OUTCOMES:
Correlation between cartilage biomarkers and Inflammatory markers | From enrollment to the end of treatment at 32 weeks
  To investigate the correlation between cartilage biomarkers (Urine CTX-II), Inflammatory markers (CBC, Ferritin, ESR, CRP) and ultrasound (HEAD-US score) comparing standard weight base low dose prophylaxis with pharmacokinetic guided extended half life FVIII concentrates

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Department, Faculty of Medicine, Chulalongkorn University and King Chulalongkorn Memorial Hospital, Bangkok, Patumwan, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 year